CLINICAL TRIAL: NCT04495998
Title: The Motor Neurological Soft Signs (MNSS) in Persons With Schizophrenia
Acronym: MNSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Susana Guimarães, MD, Principal Investigator, Faculdade de Motricidade Humana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 32/2017
Record Dates: First submitted 2020-07-25; First posted 2020-08-03 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2020-07

CONDITIONS: Psychomotor Status; Schizophrenia; Motor Skills Disorders
MeSH Terms: conditions — Status Epilepticus; Schizophrenia; Motor Skills Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motor Neurological Soft Signs (Other): motor test and an interview for the participants
  Interventions: Diagnostic Test: Brief Motor Scale_portuguese version (BMS_pt)

INTERVENTIONS:
Diagnostic Test: Brief Motor Scale_portuguese version (BMS_pt) — translate, adapt and validate Brief Motor Scale for portuguese population with schizophrenia

SUMMARY:
The aim is to contribute to the knowledge of the relationship between Motor Neurological Soft Signs (MNSS) and schizophrenia, as well as to point out the implications and recommendations for clinical and rehabilitative practices, in order to contribute to the identification of these signs as potential facilitators of prevention and a better follow-up in the psychosocial rehabilitation processes of the person with schizophrenia.

DETAILED DESCRIPTION:
The aim is to contribute to the knowledge of the relationship between Motor Neurological Soft Signs (MNSS) and schizophrenia, as well as to point out the implications and recommendations for clinical and rehabilitative practices, in order to contribute to the identification of these signs as potential facilitators of prevention and a better follow-up in the psychosocial rehabilitation processes of the person with schizophrenia.

It is therefore important to answer the following starting questions:

* How can MNSS be assessed and analysed in the Portuguese population with schizophrenia?
* How does the manifestation of MNSS differ between people with and without schizophrenia?
* Do the MNSS of people with schizophrenia vary according to their functionality level including the following areas of activity (Cognition, Mobility, Self-Care, Interpersonal Relations, Daily Activities and Participation) and their motor experiences?
* How can the information obtained by applying a validated assessment tool for this purpose be made operational as a procedure for psychomotor assessment and intervention with this population?

The following objectives have been defined to answer these questions, which guide the work:

1. Translate, adapt and validate the BMS instrument (Jahn et al., 2006) for the Portuguese population with schizophrenia;
2. Explore the relationship of MNSS with demographic variables (e.g.: age, gender, education), clinical-therapeutic variables (e.g.: age of diagnosis, number of hospitalizations, medication, type of support) and psychosocial variables (e.g.: functionality, satisfaction and well-being, motor experiences);
3. Test a multifactorial model of the relationships between MNSS, demographic variables, functional clinical-therapeutic and psychosocial;
4. Compare MNSS in people with schizophrenia and people from a healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Have a schizophrenia diagnoses

Exclusion Criteria:

* Have a motor disability
* Drugs consumer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Assessment of persons with schizophrenia with Brief Motor Scale - Portuguese version (BMS_pt) instrument | 6 weeks
  The aim of this study was to translate, adapt and validate a Portuguese version of the Brief Motor Scale (BMS_pt) in people with schizophrenia (Jahn et al, 2006).
  The participants (N=43) were evaluated twice with an interval of two weeks. In total, the sample collection lasted 6 weeks.
  Scale used and caracteristics:
  Unabbreviate title - Brief Motor Scale - Portuguese version Abbreviate title - BMS_pt Minimum value = 0; Maximum value = 2 Higher scores mean a worse outcome.
  Scale description:
  BMS_pt is a quantative test, which assessed motor neurological soft signs (MNSS) in two domains: motor coordination and motor sequencing. BMS_pt have a range score between 0 and 2 points for each item, domains and total score.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Guimarães, MD, Principal Investigator — Faculdade Motricidade Humana
Locations (1):
- Susana Guimarães, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Validity and Reliability of the Portuguese Version of Brief Motor Scale in Persons with Schizophrenia: A Preliminary Study — https://www.revistapsiquiatria.pt/index.php/sppsm/article/view/160